CLINICAL TRIAL: NCT00042406
Title: A Double-Blind, Placebo-Controlled, Randomized, Parallel Group Clinical Trial of Anti-CD4 Receptor Human Monoclonal Antibody (HuMax-CD4) in Patients With Active Rheumatoid Arthritis Failing Treatment With Methotrexate and TNF-alpha Blocking Agents
Brief Title: Trial With HuMax-CD4 in Participants With Rheumatoid Arthritis (RA) Failing Treatment With Methotrexate (MTX) and a TNF-alpha Blocker
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Hx-CD4-004
Record Dates: First submitted 2002-07-29; First posted 2002-08-01 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — zanolimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- HuMax-CD4 80 milligrams (mg) (Experimental)
  Interventions: Drug: HuMax-CD4
- HuMax-CD4 160 mg (Experimental)
  Interventions: Drug: Humax-CD4

INTERVENTIONS:
Drug: HuMax-CD4 — HuMax-CD4 80 mg was administered as a subcutaneous infusion BID with 2 weeks interval followed by administration every 4 weeks up to Week 22.
  Other Names: Zanolimumab
  Arms: HuMax-CD4 80 milligrams (mg)
Drug: Placebo — Placebo was administered as a subcutaneous infusion twice (BID) with 2 weeks interval followed by administration every 4 weeks up to Week 22.
  Arms: Placebo
Drug: Humax-CD4 — HuMax-CD4 160 mg was administered as a subcutaneous infusion BID with 2 weeks interval followed by administration every 4 weeks up to Week 22.
  Other Names: Zanolimumab
  Arms: HuMax-CD4 160 mg

SUMMARY:
The purpose of this study is to determine whether HuMax-CD4 is effective in the treatment of active RA in participants who have failed treatment with MTX and at least one TNF-alpha blocking agent.

DETAILED DESCRIPTION:
This is a multi-center, double-blind, placebo-controlled, parallel-group, randomized trial of HuMax-CD4 in the treatment of participants with active RA who have failed treatment with MTX and at least one TNF-alpha blocking agent. Participants are randomized to receive one of two doses of HuMax-CD4 or placebo. The drug will be administered as a subcutaneous infusion (given just under the skin), more often in the beginning and then followed by a maintenance dose. There is a 4 week follow up period, and the final evaluation of the clinical endpoints takes place 26 weeks after treatment start. The trial lasts about 28 weeks in all.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of rheumatoid arthritis according to the American College of Rheumatology 1987 revised criteria (ACR) of at least 6 months duration.
* Active disease at the time of screening.
* Failure to tolerate MTX, or lack of efficacy after a minimum of 6 months treatment with MTX.

Exclusion Criteria:

* Active autoimmune disease requiring therapy (other than rheumatoid arthritis and secondary Sjögren's disease).
* Syndromes such as Fibromyalgia which require chronic pain treatment.
* Most past or current cancers.
* Chronic or current infectious disease such as, but not limited to, chronic renal infection, chronic chest, nasal or throat infections, tuberculosis, hepatitis B and C.
* History of infected joint prosthesis within 5 years.
* Most active medical conditions such as heart disease, kidney disease, liver disease, blood diseases, hormonal disturbances, lung disease, psychiatric disease.
* Drug or alcohol abuse.
* Pregnant or breast-feeding women may not participate. Women of childbearing potential must use either contraceptive pills or an intra-uterine device for the entire study period.

Note: Other protocol defined Inclusion and Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2002-03-04 (Actual); Primary Completion 2003-03-31 (Actual); Study Completion 2003-03-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants with American College of Rheumatology (ACR) 20 Response | At Week 14 and Week 18
Change from Baseline in Disease Activity Score (DAS) | Baseline up to Week 26
Change from Baseline in SFP-36 questionnaire at Week 10 and 26 | Baseline, Week 10 and Week 26
Change from Baseline in C-Reactive Protein (CRP) | Baseline up to Week 26
Change from Baseline in Erythrocyte Sedimentation Rate (ESR) | Baseline up to Week 26
Number of Participants with Adverse Events (AEs) | Day 1 up to end of study (Week 26)

SECONDARY OUTCOMES:
Number of Participants With Positive Human Anti Human Antibodies (HAHA) Titres | Up to 26 weeks
Number of Participants With Clinically Significant Laboratory Abnormalities | Up to 26 weeks

CONTACTS AND LOCATIONS:
Locations (54):
- United States (50):
  - Rheumatology Associates, Montgomery, Alabama
  - Pro Health Partners, Inc., Long Beach, California
  - Rheumatology & Internal Medicine, Boling Clinical Trials, Rancho Cucamonga, California
  - Advances in Medicine, Rancho Mirage, California
  - Radiant Research, Inc., San Diego, California
  - West Coast Clinical Research, Van Nuys, California
  - Arthritis Center of CT, Waterbury, Connecticut
  - Arthritis Associates of South Florida, Delray Beach, Florida
  - Ocala Rheumatology Research Center, Ocala, Florida
  - nTouch Research, St. Petersburg, Florida
  - Radiant Research, Inc., Stuart, Florida
  - Tampa Medical Group Research, Tampa, Florida
  - nTouch Research, Decatur, Georgia
  - North Western Center for Clinical Research, Chicago, Illinois
  - Rheumatology Associates, P.C., Chicago, Illinois
  - Advocate Medical Group, Park Ridge, Illinois
  - The Arthritis Center, Springfield, Illinois
  - Deerbrook Medical Associates, Vernon Hills, Illinois
  - West Pharmaceutical Services, Evansville, Indiana
  - Idaho Arthritis & Osteoporosis Center, Meridian Hills, Indiana
  - Mercy Arthritis Center, Des Moines, Iowa
  - University of Louisville Hospital, Louisville, Kentucky
  - Osteoporosis and Clinical Trials Center, Hagerstown, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Arthritis Education and Treatment Center, Grand Rapids, Michigan
  - Midwest Arthritis Center, Kalamazoo, Michigan
  - Fiechtner Research, Lansing, Michigan
  - Westroads Medical Group, Omaha, Nebraska
  - Arthritis Center of Reno, Reno, Nevada
  - One Crouse Medical Plaza, Syracuse, New York
  - C.A.R.E. Center, Raleigh, North Carolina
  - DataPharm, Inc., Canfield, Ohio
  - Disease Study Group / Deaconess Hospital, Cincinnati, Ohio
  - Lynn Health Science, Oklahoma City, Oklahoma
  - Bend Memorial Clinic, Bend, Oregon
  - Rheumatology Clinic, Medford, Oregon
  - Providence Arthritis Center, Portland, Oregon
  - Northwest Rheumatology Associates, PC, Portland, Oregon
  - East Pennsylvania Rheumatology, Bethlehem, Pennsylvania
  - Altoona Arthritis & Osteoporosis Center, Duncansville, Pennsylvania
  - Clinical Research Center of Reading, West Reading, Pennsylvania
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - IHC Clinical Research Foundation, Salt Lake City, Utah
  - Medical College of Virginia, Div. of Rheum., Richmond, Virginia
  - Lewis Gayle Clinic, Salem, Virginia
  - Evergreen Medical & Dental Center, Kirkland, Washington
  - South Puget Sound Clinical Research Center, Olympia, Washington
  - Minor & James Med., First Hill Medical Building, Seattle, Washington
  - Internal Medicine Association of Yakima, Inc., P.S., Yakima, Washington
  - Medical Arts Center, Milwaukee, Wisconsin
- Canada (4):
  - CIADS, Medical Arts Building, Winnipeg, Manitoba
  - Ottawa Hospital-General Campus, Ottawa, Ontario
  - Sunnybrook/Women's College Research Health Science Center, Toronto, Ontario
  - Institute de Rhumtologie de Montreal, Montreal, Quebec